CLINICAL TRIAL: NCT02730715
Title: Effect of Thymoglobulin Versus Basiliximab on Regulatory T Cell Function in Live Donor Kidney Transplant Recipients
Acronym: TReg Kidney
Status: Terminated | Type: Observational
Why Stopped: Insufficient amount of T Cell collection
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 811893
Record Dates: First submitted 2016-03-24; First posted 2016-04-06 (Estimated); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: KIDNEY TRANSPLANTATION
MeSH Terms: interventions — Basiliximab; thymoglobulin; Antilymphocyte Serum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood urine and renal tissue samples (if available)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Thymoglobulin: blood specimen collection
  Interventions: Drug: Thymoglobulin
- Basiliximab: blood specimen collection
  Interventions: Drug: Basiliximab

INTERVENTIONS:
Drug: Basiliximab — Periodic blood collection to monitor Treg cells
  Other Names: Simulect
  Groups: Basiliximab
Drug: Thymoglobulin — Periodic blood collection to monitor Treg cells
  Other Names: Anti-thymocyte globulin
  Groups: Thymoglobulin

SUMMARY:
This study aims to study the effects that two standard of care immunosuppression induction regimens have on regulatory T cells (Treg) in live donor renal transplant recipients. Both regimens are currently used in this hospital for early immunosuppression induction but the effects on Treg numbers and function is not well understood and likely will impact long term immune function.

DETAILED DESCRIPTION:
This study aims to study the effects that two standard-of-care immunosuppression induction regimens have on regulatory T cells (Treg) in live donor renal transplant recipients. These two regimens use anti-T cell antibodies: thymoglobulin is a polyclonal anti-T cell preparation and basiliximab is a monoclonal anti-cluster of differentiation (CD) 25 antibody. Both are currently used in this hospital for early immunosuppression induction but the effects on Treg numbers and function is not well understood and may impact long term immune function. The investigators wish to study the effects that these standard regimens have on Treg numbers, function, and FoxP3 methylation status (an indicator of Treg function). Live donor renal transplant patients with no panel reactive antibodies (PRA) have low risk of early allograft rejection and in various transplant centers are treated with no anti-T cell immunosuppression induction or induction with thymoglobulin or basiliximab as standard of care. Most patients in this hospital receive thymoglobulin but basiliximab is used as well. There are no proven long term benefits to either approach but each seems to lower the risk of short term acute cellular rejection. Both of these agents have been shown to affect numbers of Tregs (as they are T cell subsets) but data does not exist on the duration of these effects or the effects that these agents have on Treg potency or Treg FoxP3 methylation status. Since Tregs are believed to be important in long term control of immune responses, it is possible that the reason these agents do not improve long term results in spite of their short term improvement in rejection rate is due to effects on Treg.

T cell depletion by antibody has become standard of care in the majority of renal transplant programs in the country (including Penn) and this may have reduced short term acute rejection episodes within the first year of transplant. There have unfortunately not been corresponding improvements in long term outcomes and, in fact, the average half life of a renal graft is minimally changed in 2010 compared to 1995. This has been attributed to unresolved issues in diagnosing and treating what is described as "chronic allograft nephropathy" - which in real terms, is probably a longstanding chronic rejection that may be in part due to a mixed T and B cell antigraft response. Despite the fact that these agents are used regularly in clinical transplantation, little is known about their effects on regulatory T cell (Treg) numbers and suppressive activity and nothing is known about effects on the methylation status of Tregs, which seems to correlate with their function. These are novel questions that are a) relevant to clinical practice since these agents are being used in renal transplantation already, b) may yield information that could alter best practices, and c) will yield more basic information about Tregs in human transplantation that will be relevant to future study. There have been few papers that have looked predominantly at a few immunosuppressive agents and numbers of Tregs (this is a low quality statistic since the markers of Tregs are shared by other cell types and thus the "numbers" can be hard to interpret) but little about function or methylation. The investigators propose to randomize 30 live donor kidney recipients to receive either thymoglobulin or basiliximab immunosuppression and thereafter receive standard of care maintenance immunosuppression determined by the clinical team. Both of these regimens are used as standard of care in this hospital. The investigators will enroll only patients with low immunological risk (0-10% PRA) and who are receiving an Blood Type (ABO) compatible transplant. After the initial randomization, all further decisions regarding immunosuppression will be made by the clinical team independent of the study. The investigators will draw blood samples pre-transplant, 3 months after transplant, and 6 months and 12 months after transplant.

ELIGIBILITY:
Inclusion Criteria:

* adult patients receiving first live donor kidney transplant. 0-10% panel reactive antibody

Exclusion Criteria:

* HIV positive, hepatitis C positive, pregnancy, inability to provide informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Live donor renal transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2010-11 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Absolute Treg number Cells | 5 years
  Each sample will be measured by flow cytometry. Data will be analyzed for each treatment arm using nonparametric statistical tests and expressed as the medium value and inter-quartile range.
Treg function tested by flow cytometry. | 5 years
  T cells and Tregs will be isolated. T cells will be labeled with CFSE and induced to proliferate by addition of CD3 mAb. Data will be evaluated by nonparametric methods.

SECONDARY OUTCOMES:
Treg methylation | 5 years
  An indicator of Treg function will be determined by purifying Tregs and monitoring methylation after bisulphate conversion and DNA sequencing. Percentages of methylated CpG sites/samples and will be compared by nonparametric statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew L Levine, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States